CLINICAL TRIAL: NCT03868397
Title: Preoperative Portal and Splanchnic Flow Measurement in Living Donor Liver Transplantation Recipient With Spontaneous Portosystemic Shunt at MRI: Preliminary Study
Brief Title: Preoperative Portal and Splanchnic Flow Measurement Using MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Hee Yoon, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SNUH-2017-1262
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Liver Cirrhoses
Keywords: MRI; cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver MRI (Experimental): In this study, MRI refers to phase-contrast 4D flow sequence.
  Interventions: Diagnostic Test: Liver MRI

INTERVENTIONS:
Diagnostic Test: Liver MRI — Liver MRI including 4D flow sequence is performed twice in liver transplantation recipients, before and 1 month-after transplantation.
  In donor candidates, liver MRI including 4D flow sequence is performed twice in 1-3 weeks to assess repeatability of the technique.

SUMMARY:
This study aims to assess the alteration of portal and splanchnic flow using MRI after liver transplantation in patients with splenomegaly or splenic varix.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* And signed informed consent
* And planned either a) liver transplantation as a recipient; or b) liver transplantation as a donor

Exclusion Criteria:

* any absolute/relative contraindication of contrast-enhanced MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Portal flow | in a month after 2nd MRI
  portal flow measured with MRI (4D flow sequence)

SECONDARY OUTCOMES:
SMV flow | in a month after 2nd MRI
  superior mesenteric vein (SMV) flow measured with MRI (4D flow sequence)
Splenic vein flow | in a month after 2nd MRI
  splenic vein flow measured with MRI (4D flow sequence)
splenic varix flow | in a month after 2nd MRI
  splenic varix flow measured with MRI (4D flow sequence) only in liver recipients

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hee Yoon, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No